CLINICAL TRIAL: NCT01690000
Title: Treatment of Osteopenia With Melatonin: Effects on BMD, Muscle Strength and Quality of Life
Brief Title: Treatment of Osteopenia With Melatonin
Acronym: MelaOst
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2011-AKA
Record Dates: First submitted 2012-06-28; First posted 2012-09-21 (Estimated); Results first posted 2016-05-06 (Estimated); Last update posted 2016-05-06 (Estimated); Status verified 2013-04

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis | interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Melatonin1 (Active Comparator): 1 mg melatonin nightly
  Interventions: Drug: Melatonin
- Melatonin3 (Active Comparator): 3 mg melatonin given nightly
  Interventions: Drug: Melatonin
- Placebo (Active Comparator): Identical placebo given nightly
  Interventions: Drug: Melatonin

INTERVENTIONS:
Drug: Melatonin — 1 or 3 mg of melatonin PO each night for 12 months

SUMMARY:
The aim of the study is to assess the effect of melatonin treatment in patients with osteopenia on BMD, muscle function, quality of life and calcium homeostasis.

DETAILED DESCRIPTION:
Background: Melatonin is known for its regulation of circadian rhythm. The production falls with age, which explains why elderly may have disturbed sleep patterns. Laboratory study and animal experimental studies suggests that melatonin also may protect against bone loss through increased osteoblast- and inhibited osteoclast activity. However, so far human studies have not been performed.

Design and patients: Double blinded randomised controlled study. Eighty post-menopausal women (aged 55-75) with osteopenia are randomized to receive 1mg, 3mg or placebo (daily - at night time) for 12 months.

Methods and results: Effects of melatonin on BMD, bone- structure and mass will be assessed through DXA-scans, pQCT, and QCT. Quality of life, sleep, and activity level will be assessed though questionnaires. Calcium homeostasis will be analyzed through blood and urines samples. As safety parameters, balance and muscle function will also be performed.

Conclusion: Expected improvements in BMD, quality of life and sleep.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women between 55 and 75 years.
* Osteopenia verified by DXA-scans of total hip or lumbar spine (t-score between -1 and -2.5)
* Written informed consent after oral and written information

Exclusion Criteria:

* Severely impaired renal function (plasma creatinine >60 eGFR ml/l).
* Severely impaired hepatic function (Plasma alanine aminotransferase (ALAT) and/or alkaline phosphatase more the doubled compared to upper limit of reference value).
* Coagulation factors PP <0.6
* Hypercalcemia (p-ion calcium > 1.32 nmol/l)
* Previous or present malignancies (except a treated skin cancer that is not melanoma or treated carcinoma in situ, 2 years since last therapy).
* Diseases affecting the calcium homeostasis including untreated thyroid diseases.
* Regular use of medicine affecting the calcium homeostasis; including diuretics, lithium, antiepileptica, glucosteroids.
* SSRI-product with fluvoxamin.
* Treatment with carbamazepin
* Treatment with rifampicin
* Severe malabsorption syndrome including gastric or intestinal resection.
* Alcohol or drug abuse.
* Smokers
* Major medical or social problems that will be likely to preclude participation for one year.

Ages: 55 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2012-11; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anne Kristine Amstrup, MD, Principal Investigator — Osteoporoseklinikken, Dept. of Endocrinology and Internal Medicine (MEA) Aarhus University Hospital, Tage-Hansens Gade 2, AArhus, DEnmark
Locations (1):
- Osteoporoseklinikken, dept of Endocrinology and Internal Medicine (MEA), Aarhus C, Denmark

REFERENCES:
- [Derived] Amstrup AK, Sikjaer T, Mosekilde L, Rejnmark L. The effect of melatonin treatment on postural stability, muscle strength, and quality of life and sleep in postmenopausal women: a randomized controlled trial. Nutr J. 2015 Sep 30;14:102. doi: 10.1186/s12937-015-0093-1. PMID 26424587

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We recruited 81 postmenopausal women with osteopenia to receive either melatonin (n=40) (1 or 3 mg) or similar placebo (n=41) nightly for 12 months. In addition, all women received a daily supplementation with 800mg calcium and 20ug D3
Pre-assignment Details: A total of 202 women were invited to participate. 81 were included in the study
Groups:
- Melatonin1+3: Melatonin: 1 or 3 mg of melatonin PO each night for 12 months
- Placebo: Identical placebo given nightly for 12 months
Period: Overall Study
Arm/Group | Melatonin1+3 | Placebo
Started | 40 | 41
Completed | 37 | 35
Not Completed | 3 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Melatonin1+3 | Placebo | Total
Number analyzed (Participants) | 40 | 41 | 81
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 32 | 29 | 61
  >=65 years | 8 | 12 | 20
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 41 | 81
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Denmark | 40 | 41 | 81

OUTCOME MEASURES:

1. Primary Outcome: Changes in Bone Mineral Density (BMD)
Description: Effects of melatonin on BMD will be assessed through DXA-scans
Time Frame: baseline and end of study (after 12 months)
Measure: Mean (Standard Error); unit: percentage of change in BMD
Groups:
- Melatonin1+3: 1+3 mg melatonin nightly
  Melatonin: 1 or 3 mg of melatonin PO each night for 12 months
Arm/Group | Melatonin1+3 | Placebo
Number analyzed (Participants) | 39 | 37
percentage of change in BMD | -0.05 (3.07) | -1.45 (2.81)
Statistical Analysis 1: Comparison: Melatonin1+3 vs Placebo; The p-value was calculated; Test type: Superiority or Other; p < 0.05, t-test, 2 sided — The p-value was calculated

2. Secondary Outcome: Changes in Calcium Homeostasis
Description: Calcium homeostasis will be analyzed through blood and urines samples
Time Frame: baseline, after 3, 6, 9 months, and end of study (after 12 months)
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 12 months (entire study period)
Arm/Group | Melatonin1+3 | Placebo
Serious Adverse Events (participants affected / at risk) | 5/40 | 7/41
Other Adverse Events (participants affected / at risk) | 19/40 | 17/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Melatonin1+3 (N=40) | Placebo (N=41)
Planned operation (Musculoskeletal and connective tissue disorders) | 5 (5) | 7 (7) — Pre-planned operation of known musculoskeletal or cardiac complaints not related to the study.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Melatonin1+3 (N=40) | Placebo (N=41)
Infection not assumed related to study medicine (Infections and infestations) | 19 (22) | 17 (21)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No